CLINICAL TRIAL: NCT06681792
Title: The Effect of Climate Change Workshops Based on Protection Motivation Theory on Primary School Students' Climate Change Awareness, Environmental Awareness and Eco-Friendly Behaviors: a Randomized Controlled Trial
Brief Title: Workshops Based on Protection Motivation Theory and Climate Change
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Deniz Kocoglu-Tanyer, Prof.Dr, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/50
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Health Behavior; Climate Change; Students
Keywords: Protection Motivation Theory; Primary School Students; Climate Change; Awareness; Eco-friendly behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking will not be possible due to the method of application of this study. However, the data collector, statistician and reporting will be masked during the research process. In the research process, pre-test data will be collected by the teachers workin in the study school. The post-test data will be collected by another researcher (a researcher trained in the data collection form and trained in the field of nursing). The research data will be transferred to the computer by the researcher who collected the post-test data by coding the experimental and control groups as 'environment' and 'world' respectively. The transferred database will be analysed by a statistical expert. After the research report has been written, the codings made for the experimental and control groups will be explained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The experimental group will take part in seven weekly workshops based on Protection Motivation Theory .
  Interventions: Behavioral: Climate Change Workshops Based on Protection Motivation Theory
- Control Group (No Intervention): The control group will not receive any intervention. It was planned to apply the data collection instruments to the control group under the supervision of the researcher and in parallel with the intervention group during the same period.

INTERVENTIONS:
Behavioral: Climate Change Workshops Based on Protection Motivation Theory — The experimental group will take part in seven weekly workshops. One workshop will last 40 minutes.The workshop to be applied to the experimental group will take place every week and will last 40 minutes. The workshops, which are based on the Protection Motivation Theory, consist of topics such as the balance of nature, climate change, carbon and ecological footprints, reducing the effects of climate change and adaptation workshop, acquiring environmentally friendly behaviour, recycling and the Green School Programme for sustainable environmental education.
  The workshops include interactive applications such as students expressing their thoughts on the weekly themes, games, brainstorming, word cloud, planting trees, painting cloth bags, watching videos, making presentations on the themes. Motivation Theory, consist of topics such as the balance of nature, climate change, carbon and ecological footprints, reducing the effects of climate change and adaptation workshop, acquiring enviro
  Arms: Intervention Group

SUMMARY:
The research will be conducted to determine the effect of climate change workshops based on the Protection Motivation Theory on students' climate change awareness, environmental awareness and environmentally friendly behaviours. The aim of this study is to develop climate change awareness, environmental awareness and sustainable behavioural change in primary school students to cope with climate change by adopting eco-friendly behaviours.

DETAILED DESCRIPTION:
Climate change is a global problem and one of the most important public health issues of the 21st century. The direct and indirect impacts of climate change on human health are as follows. While it poses unique and significant threats to public health and well-being through direct impacts on heat stress, flooding and the spread of infectious diseases, food and water insecurity, conflict and migration, and in relation to fossil fuels, it also adversely affects human health through indirect impacts on livelihoods, equity, community health and social support structures, which are social determinants of health.

Due to the increasing effects of climate change, many different disciplines such as physics, biology, meteorology and geology are carrying out important studies with the main aim of halting the negative trend and ensuring the survival of species. In addition to scientific studies, many institutions and organisations are raising awareness of climate change and encouraging people to take institutional and individual action. Scientific studies in the field of health focus on understanding the effects of climate change on human health and evaluating the impact of interventions that focus on individual behaviour change in the fight against climate change. These are interventions such as sending messages for environmentally friendly behaviour, online chats, nature-based education programmes, watching films and peer education.

When the effectiveness of these interventions is evaluated, it is seen that they have a positive effect in reducing the negative consequences of climate change while improving their environmental knowledge, attitudes and intentions. However, while the impact of the interventions on climate change is small while the interventions are ongoing, there is no evidence of a positive impact when the interventions end. The fact that the effects of interventions are long-lasting highlights the need for interventions that are modelled and targeted at younger age groups to achieve behaviour change. The theory of protective motivation, which is based on the assessment of the magnitude of harm caused by an event, the likelihood of the event occurring and the presence of a protective activity, is a promising theory for mitigating the impacts of climate change and achieving behaviour change.

This theory, which is educational and motivational, offers suggestions as to why people tend to engage in unhealthy practices and how these behaviours can be changed. From the literature, it is known that interventions with primary school children can lead to recycling awareness, environmental sensitivity, eco-donation and eco-action. In order for these effects to be lasting, it is also important to ensure the permanence of threat awareness and coping. For this reason, this study examines the effect of climate change workshops based on Protection Motivation Theory for primary school students on the outcomes of students' environmental awareness, climate change awareness and adoption of environmentally friendly behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Being 9-10 years old and attend the school where the study is being conducted,
* Voluntarily agree to take part in the research,
* Consent from the student's family to participate in the study,

Exclusion Criteria:

* If the pupil has an allergy to plants or grass

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Climate change awareness | T0 (Pre-test) T1 (15 days after the end of the procedure) T2 (3 months after the end of the procedure)
  Knowledge about the definition, causes and consequences of climate change. It has included three questions.
  * Marking the sentences related to the definition of climate change as true/false
  * Identify the causes of climate change among the options
  * Finding the consequences of climate change among the options
The Scale of Attitude Towards the Environment | T0 (Pre-test) T1 (15 days after the end of the procedure) T2 (3 months after the end of the procedure)
  The scale developed by Peker and Ceylan (2020) consists of three sub-dimensions and 15 items. The reliability coefficient (Cronbach's alpha) of the scale was found to be 0.871. The Kaiser-Mayer-Olkin test of the scale was 0.877; Barlett's test was 1623.380 (p<0.01). The sub-dimensions of the scale were grouped as pollution, love of animals and love of plants and nature. The Cronbach's alpha values of the sub-dimensions are 0.853, 0.723 and 0.674 respectively. The items are measured on a three-point Likert scale (1: disagree, 2: partly agree, 3: agree). An increase in the score indicates a positive attitude.
Eco-friendly behaviours | T0 (Pre-test) T1 (15 days after the end of the procedure) T2 (3 months after the end of the procedure)
  The measure will be the number of implementations by students of 23 environmentally friendly behaviours defined on the basis of literature.

SECONDARY OUTCOMES:
The Questionnaire on Children's Perceptions of the Four Elements of the Theory of Protective Motivation | T0 (Pre-test) T1 (15 days after the end of the procedure) T2 (3 months after the end of the procedure)
  This questionnaire assesses students' agreement with 9 statements assessing the concepts of perceived threat sensitivity(2) , perceived threat severity (2), perceived response effectiveness (3) and self-efficacy (2)in relation to the climate crisis. For each proposition there are options of agree (3), undecided (2) and disagree (1). It was developed based on the literature related to the model and evaluated by experts. This form is used to assess change situation for each concept. An increase in the score is indicative of an enhanced perception of the situation in question.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuvayi Milli İlkokulu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data supporting this study are not publicly available due to ethical reasons but the datasets used and/or analyzed during the current study are available by emailing deniizkocoglu@gmail.com upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 2 years after the publication of results
Access Criteria: the datasets used and/or analyzed during the current study are available by emailing deniizkocoglu@gmail.com upon reasonable request.